CLINICAL TRIAL: NCT01816399
Title: Spacial Relation of QRS-T Vectocardiogram is a Good Predictor of Coronary Disease in Patients With Normal Rest 12-leads ECG
Brief Title: New Vectorcardiogram Analysis a Good Predictor of Coronary Disease in Patients With Normal Rest 12-leads ECG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-9-2003b
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Routine coronary angiography patients
  Interventions: Procedure: Routine coronary angiography

INTERVENTIONS:
Procedure: Routine coronary angiography

SUMMARY:
The aim of this study is to determine whether a new vectorcardiogram (VCG) analysis will facilitate the detection of significant coronary disease (CAD) in patients with normal rest 12-leads ECG (NE).

DETAILED DESCRIPTION:
Patients with NE will undergo coronary angiography for routine indications. Prior to the angiography a computerized simultaneous multi-leads ECG will be recorded and, using a new dedicated algorithm for 3D electrical activity reconstruction, the investigators will plot the horizontal VCG of the whole ECG cycle. Using this new VCG analysis we will determine whether the patients have normal coronary arteries or coronary disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with normal rest 12-leads ECG

Exclusion Criteria:

* Patients with significant irregular heart beat
* Patients with heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing routine coronary angiography
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Detection of CAD in patients undergoing routine coronary angiography | One month
  Following angiography patients will be categorized as having normal coronary arteries (NC) or coronary disease (CD) if more than 50% lumen diameter narrowing is found in one of the arteries.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel